CLINICAL TRIAL: NCT01465568
Title: Denosumab in Current Users of Bisphosphonates for Glucocorticoid-induced Osteoporosis: a Randomized Controlled Trial
Brief Title: Denosumab in Current Users of Bisphosphonates for Glucocorticoid-induced Osteoporosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tuen Mun Hospital (Other Government)
Responsible Party: Principal Investigator, Chi Chiu Mok, Consultant, Tuen Mun Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CREC/984/11
Record Dates: First submitted 2011-10-30; First posted 2011-11-07 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Osteoporosis
Keywords: osteoporosis; denosumab; RANKL; glucocorticoids
MeSH Terms: conditions — Osteoporosis | interventions — Denosumab; Diphosphonates

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Denosumab (Active Comparator): denosumab
  Interventions: Drug: Denosumab
- bisphosphonates (Active Comparator): continuation of bisphosphonates
  Interventions: Drug: bisphosphonates

INTERVENTIONS:
Drug: Denosumab — 60mg subcutaneous injection 6 monthly for 2 doses
  Other Names: Prolia
  Arms: Denosumab
Drug: bisphosphonates — continue present bisphosphonate treatment
  Other Names: continuation of bisphosphonates in their usual dosages
  Arms: bisphosphonates

SUMMARY:
The purpose of this study is to study the efficacy of denosumab, a new drug, in the treatment of osteoporosis in patients using bisphosphonates.

DETAILED DESCRIPTION:
There are no data on the use of denosumab in steroid induced osteoporosis. Postmenopausal women with chronic use of Glucocorticoid (GCs) are at high-risk of osteoporotic fractures. Despite bisphosphonate treatment, a certain proportion of high-risk patients using chronic GCs either do not achieve a satisfactory gain in bone mineral density (BMD) or develop new fragility fractures. Thus, more potent osteoporosis treatment is necessary for this subgroup of patients. This prompts the current study which aims to examine the efficacy of denosumab in current users of oral bisphosphonates for Glucocorticoid-induced Osteoporosis (GIOP).

ELIGIBILITY:
Inclusion Criteria:

1. Women or adult men (>18 years of age) with various medical diseases requiring long-term prednisolone treatment. Pre-menopausal women should have no plan for pregnancy within 2 years of study entry and agree to practice contraception during this 2-year period.
2. A daily dose of prednisolone (or equivalent) of more than 2.5mg within 3 months of study entry.
3. Having received oral bisphosphonate treatment for at least 2 years.
4. Suboptimal response to bisphosphonate treatment, defined as either one of the following: (1) failure of lumbar spine, femoral neck or total hip BMD values to increase; (2) values of lumbar spine, femoral neck or total hip BMD remain osteoporotic, ie. T scores < -2.5 or Z scores < -2.0; or (3) development of new fragility vertebral or non-vertebral fractures despite at least 2 years' treatment with good compliance.
5. Informed consent from patients.

Exclusion Criteria:

1. Patients with previous use of denosumab or teriparatide.
2. Premenopausal women who plan for pregnancy within 2 years of study entry or who do not agree for contraception within this 2-year period.
3. Patients with known bone disorders such as osteomalacia, renal osteodystrophy, and hyperparathyroidism.
4. Patients with unexplained hypocalcemia.
5. Patients with serum creatinine level of >=200umol/L.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-12; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
bone mineral density (BMD) changes at the lumbar spine | baseline, 6 months and 12 months

SECONDARY OUTCOMES:
BMD changes in the total hip and femoral neck | baseline, 6 months and 12 months
bone turnover markers | baseline, 6 months and 12 months
New vertebral fractures | 12 months
adverse events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Chi Chiu Mok, MD, FRCP, Principal Investigator — Tuen Mun Hospital
Locations (1):
- Tuen Mun Hospital, Hong Kong, China

REFERENCES:
- [Derived] Mok CC, Ho LY, Ma KM. Switching of oral bisphosphonates to denosumab in chronic glucocorticoid users: a 12-month randomized controlled trial. Bone. 2015 Jun;75:222-8. doi: 10.1016/j.bone.2015.03.002. Epub 2015 Mar 8. PMID 25761434